CLINICAL TRIAL: NCT04433130
Title: Eye Health in Children and Adolescents: Repeated Cross-sectional Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Sun Yat-sen University (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: SYSU-OPH-006
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator will take a mixed-methods approach to gather relevant information from both children or adolescents, and their parents on profiles of eye health, as well as routinely available indicators. This includes a series of baselining and follow-up analyses of cohort data collected on epidemiological, clinical, therapeutic, and service aspects of eye health and individual-level outcomes

DETAILED DESCRIPTION:
The investigator will take a mixed-methods approach to gather relevant information from both children or adolescents, and their parents on profiles of eye health, as well as routinely available indicators. This includes a series of baselining and follow-up analyses of cohort data collected on epidemiological, clinical, therapeutic, and service aspects of eye health (e.g., social environment, preventive behaviours, risk factors, knowledge and attitudes, health and social care, etc.) and individual-level outcomes (e.g., clinical parameters and symptoms, biomarkers, self-reported measures, risk profiles, etc.).

ELIGIBILITY:
Inclusion:

* Subjects with valid information on eye health-related profiles
* Completion of eye health examination delivered by trained ophthalmic professionals

Exclusion:

* Inability to give informed consent
* Unable to retrieve individual records on eye health examination

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects seeking care on refractive error or vision problems and their parents
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
visual acuity | Baseline and changes up to 4 years
  The primary aims of the research project are to explore the profiles of eye health and how lifestyle behaviours, social environment, and individual risk factors are associated with health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China